CLINICAL TRIAL: NCT04353661
Title: ¹²⁹XE MRI Assessment Of Disease Progression In Patients With Chronic Obstructive Pulmonary Disease Treated With Standard-of-Care Medications With Or Without Daily Open-Label Azithromycin Treatment To Prevent Acute Exacerbation
Brief Title: A Study Of ¹²⁹XE MRI To Assess Disease Progression In Patients With COPD Treated With Or Without Azithromycin And Standard-of-Care Medications
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated by Sponsor due to patient recruitment challenges.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE42063
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label, parallel group, randomized controlled trial (RCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A Open-label: azithromycin + SOC therapy (Experimental): Participants will receive azithromycin and SOC theraphy for 52 weeks.
  Interventions: Drug: Azithromycin; Other: HP xenon (¹²⁹XE)
- Arm A Open-label: SOC therapy (Active Comparator): Participants will receive SOC theraphy for 52 weeks.
  Interventions: Other: HP xenon (¹²⁹XE)
- Arm B Observational: SOC therapy (Active Comparator): Participants will receive SOC theraphy for 52 weeks.
  Interventions: Other: HP xenon (¹²⁹XE)

INTERVENTIONS:
Drug: Azithromycin — Azithromycin will be administered orally.
  Arms: Arm A Open-label: azithromycin + SOC therapy
Other: HP xenon (¹²⁹XE) — HP xenon (¹²⁹XE) will be administered at specified timepoints and the total dose bag volume should target 20% of the patient's forced vital capacity followed by a breath hold of up to 15 seconds

SUMMARY:
This study will test whether daily use of azithromycin will reduce the rate of exacerbations and improve lung ventilation and perfusion assessed by XE-MRI. The sensitivity of XE-MRI to detect COPD progression will be compared with standard clinical assessment measures including standard lung function tests, 6 minute walk test, and patient reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smokers with years ≥ 10 pack years
* mMRC dyspnea score > 1
* Post-bronchodilator FEV-1/forced vital capacity (FVC) <0.70 at Visit 1 or Visit 2
* Cohort A: GOLD Stage 2-4 COPD with a history of ≥ 2 moderate/severe exacerbations within a 12-month period in the 24 months prior to screening
* Cohort B: GOLD Stage 1 COPD with a history of ≥1 moderate/severe exacerbations within a 12-month period in the 24 months prior to screening
* Receiving SOC background drug therapy as per GOLD or British Thoracic Society (BTS) guidance for COPD for 12 weeks prior to screening Visit 1
* On an eligible bronchodilator medication (LABA ± LAMA) ± ICS therapy for ≥12 weeks prior to Visit 1
* Chest X-ray or CT scan within 6 months prior to Visit 1, or during the screening period (prior to Visit 2), that confirms the absence of clinically significant lung disease besides COPD
* Use of contraceptive measures

Exclusion Criteria:

* Diagnosis of significant respiratory disease other than COPD
* Comorbid conditions that may interfere with the evaluation of an investigational medical product
* Known sensitivity or allergy to azithromycin
* A COPD exacerbation and or pneumonia within 4 weeks prior to Visit 1
* Use of systemic corticosteroids within 4 weeks (oral or intravenous) or within 12 weeks (intramuscular IM) prior to screening Visit 1
* MRI is contraindicated
* Any known arrhythmia, bradycardia or severe cardiac insufficiency
* Participant can not hold breath for 15 seconds
* Participant does not fit in the ¹²⁹XE vest coil used for MRI
* Pregnant, lactating, or intending to become pregnant during the study or within 4 weeks after the last dose of the investigational medical product
* History or evidence of substance abuse that would pose a risk to participants safety, interfere with the conduct of the study, or have an impact on the study results
* For participants in Cohort A: Known significant hearing impairment as indicated by a score of ≥ 26 on the Hearing Handicap Inventory in the Elderly-Screening Questionnaire or as determined by the investigator
* History of Clostridium difficile (C. difficile) diarrhea Clinically significant ECG changes, which in the opinion of investigator warrants further investigation or with a QTc interval > 450 ms

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genetech
Locations (2):
- United States (2):
  - Duke Asthma Allergy and Airway Center, Durham, North Carolina
  - University of Virginia Health System, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Open-label: Azithromycin + SOC Therapy: Participants received azithromycin and SOC therapy for 52 weeks.
- Arm A Open-label: SOC Therapy; Arm B Observational: SOC Therapy: Participants received SOC therapy for 52 weeks.
Period: Overall Study
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational: SOC Therapy
Started | 3 | 5 | 4
Completed | 2 | 4 | 2
Not Completed | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Study termination by the Sponsor | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational: SOC Therapy | Total
Number analyzed (Participants) | 3 | 5 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 6
  >=65 years | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 3 | 4 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in 129Xenon (129Xe) Magnetic Resonance Imaging (MRI) Ventilation Defect Percentage (VDP) From Baseline to Week 24
Description: Hyperpolarized 129Xe gas was administered to the participants at specified timepoints. MRI using hyperpolarized 129Xe was used for 3D mapping of ventilation and gas distribution in the alveolar space and its uptake in interstitial barrier tissues as well as its transfer to red blood cells. Positive change from baseline indicated worse outcomes.
Time Frame: Baseline up to Week 24
Population: ITT population. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: ventilation defect percentage
Groups:
- Arm B Observational : SOC Therapy: Participants received SOC therapy for 52 weeks.
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational : SOC Therapy
Number analyzed (Participants) | 3 | 4 | 2
ventilation defect percentage | 6.33 (12.70) | -1.75 (5.12) | -1.00 (7.07)

2. Secondary Outcome: Number of Participants With Adverse Events (AE) With Severity Determined According To The World Health Organization (WHO) Toxicity Scale
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptoms, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. The WHO toxicity grading scale was used for assessing adverse event severity. Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening; Grade 5: death. There were no participants with grade 5 AEs. Participants were counted once at their highest AE reported.
Time Frame: Baseline up to Week 52
Population: Safety population
Measure: Number; unit: Number of Participants
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational: SOC Therapy
Number analyzed (Participants) | 3 | 5 | 4
Number of Participants
  Grade 1 | 0 | 1 | 0
  Grade 2 | 1 | 1 | 1
  Grade 3 | 1 | 1 | 1
  Grade 4 | 1 | 2 | 1

3. Secondary Outcome: Change in 129Xe MRI VDP From Baseline to Week 48
Description: as for outcome 1
Time Frame: Baseline to Week 48
Population: ITT Population. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: ventilation defect percentage
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational: SOC Therapy
Number analyzed (Participants) | 2 | 3 | 3
ventilation defect percentage | 0.50 (6.36) | -6.00 (9.85) | -4.67 (7.77)

4. Secondary Outcome: Change in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1, Liters) From Baseline to Week 24 and Week 48
Description: FEV1 is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration. Positive change from baseline indicated better outcomes.
Time Frame: Baseline to Week 24 and Week 48
Population: ITT Population. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational: SOC Therapy
Number analyzed (Participants) | 1 | 2 | 2
liters
  Change from Baseline at Week 24 | 0.15 (NA) — The standard deviation was not estimable for a single participant. | -0.01 (0.21) | -0.12 (0.04)
  Change from Baseline at Week 48 | 0.19 (NA) — The standard deviation was not estimable for a single participant. | -0.03 (0.17) | -0.26 (0.14)

5. Primary Outcome: Rate of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Over 48 Weeks
Description: A moderate COPD exacerbation was defined as new or increased COPD symptoms (e.g., dyspnea, sputum volume, and sputum purulence) for at least 2 consecutive days that led to treatment with systemic corticosteroids and/or antibiotics. A severe COPD exacerbation was defined as new or increased COPD symptoms (e.g., dyspnea, sputum volume, and sputum purulence) for at least 2 consecutive days that led to hospitalization or death.
Time Frame: Baseline up to Week 48
Population: ITT population
Measure: Mean (Standard Deviation); unit: exacerbations per year
Arm/Group | Arm A Open-label: Azithromycin + SOC Therapy | Arm A Open-label: SOC Therapy | Arm B Observational : SOC Therapy
Number analyzed (Participants) | 3 | 5 | 4
exacerbations per year | 1.41 (1.70) | 1.06 (1.11) | 0.23 (0.47)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 48
Groups:
- Cohort A - SOC + Azithromycin: Participants received azithromycin and SOC theraphy for 52 weeks.
- Cohort A - SOC; Cohort B - SOC: Participants received SOC theraphy for 52 weeks
Arm/Group | Cohort A - SOC + Azithromycin | Cohort A - SOC | Cohort B - SOC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 2/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - SOC + Azithromycin (N=3) | Cohort A - SOC (N=5) | Cohort B - SOC (N=4)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - SOC + Azithromycin (N=3) | Cohort A - SOC (N=5) | Cohort B - SOC (N=4)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT04353661/Prot_SAP_000.pdf